CLINICAL TRIAL: NCT03915327
Title: Short-term Use of Intravenous Iron Isomaltose Anhydride for Preoperative Anemic Patients Undergoing Orthopedic Surgery: a Prospective, Randomized, Controlled Study
Brief Title: Short-term Intravenous Iron Isomaltose Anhydride for IDA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Associate Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCH20190308
Record Dates: First submitted 2019-03-31; First posted 2019-04-16 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron-deficiency anemia; Intravenous iron isomaltose anhydride; Preoperative
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous iron group (Experimental): Enrolled subjects would receive intravenous iron isomaltose anhydride within 24 hours of the subject's inclusion.
  Interventions: Drug: Intravenous iron isomaltose anhydride
- Control group (No Intervention): Clinical management, including surgical procedures, anesthesia, and perioperative management, are performed in accordance with standard clinical practice.

INTERVENTIONS:
Drug: Intravenous iron isomaltose anhydride — Enrolled subjects would receive intravenous iron isomaltose anhydride within 24 hours of the subject's inclusion.
  Arms: Intravenous iron group

SUMMARY:
This prospective, randomized, controlled study aims to evaluate the impact of short-term intravenous iron isomaltose anhydride on postoperative recovery and the requirement for allogeneic red blood cells (RBC) transfusion in preoperative Iron-deficiency anemia (IDA) patients receiving orthopedic surgery, thus facilitating developing a simple and effective iron supplement approach for patients' recovery.

DETAILED DESCRIPTION:
Anemia is a decrease in the concentration of hemoglobin (Hb) or RBC count in the blood ting, causing body not being able to adequately supply oxygen to tissues and cells. Preoperative anemia is common in patients receiving elective surgery, with a prevalence ranging from 5% to 75%. For instance, the prevalence of anemia before total hip or total knee arthroplasty is around 35%. Preoperative anemia is one of the main predictors of perioperative allogeneic RBC transfusion, and is closely associated with postoperative infection, increased morbidity and mortality, prolonged hospital stay, and decreased quality of life.

As the world enters an aging society, the proportion of elderly patients receiving surgery, especially orthopedic surgery, is increasing. There are 3 main causes of anemia in the elderly: nutritional anemia (~34%), which is caused by lack of hematopoietic materials. Iron-deficiency anemia (IDA) is the most common type of nutritional anemia, while megaloblastic anemia caused by lack of folic acid and vitamin B12 is relatively rare. Anemia of chronic disease (~32%), which is characterized by disorders of iron metabolism that occurs in certain chronic diseases, such as persistent infections, inflammation and tumors. Anemia of unknown cause (-34%), which may involve multifactorial pathogenic mechanisms and comorbidities. IDA, the most common cause of perioperative anemia in patients receiving orthopedic surgery, is a condition caused by hematopoietic materials deficiency and has a good clinical response to iron supplementation with a rapid rise of Hb level. Iron supplementation in patients with preoperative IDA, or insufficient iron intake and excessive loss is able to improve the patients' surgical tolerance and reduce the transfusion rate; For anemic patients with acute blood loss during surgery, iron supplementation is able to accelerate anemia correction, thus enhancing postoperative recovery and shortening length of hospital stay.

Iron therapy can be administrated by the oral or intravenous route. Absorption of oral iron therapy is relatively low, and it usually takes over 1 to 2 months to correct the iron deficiency status. Therefore, intravenous iron therapy is recommended for patients diagnosed with IDA after admission to hospital to receive surgery. Intravenous iron therapy was originally the standard iron supplementation in chronic renal failure patients with IDA. Subsequently, it was expanded to the anemia of patients with conventional inflammatory bowel disease for its desirable efficacy. Several studies of elderly IDA patients receiving orthopedic surgery and gynecologic surgery suggest that intravenous iron therapy can rapidly increase hemoglobin levels before surgery, leading to a decrease in blood transfusion rates. The calculation of the total dose of intravenous iron is as follows:

= Weight (kg) ×[Target Hb level（g/L）- actual Hb level（g/L）] ×0.24 + 500mg Treatment duration is over 2 weeks in most clinical studies of intravenous iron therapy. In China, few patients are treated with intravenous iron therapy in community hospitals for 2 to 4 weeks before surgery. Therefore, many IDA patients did not receive proper preoperative intravenous iron therapy. Iron isomaltose anhydride, an intravenous iron preparation that can be administered in a single treatment up to 1000 mg in a relatively short (15 minutes) time without need for test dose, is of low risk of adverse reactions. Therefore, sufficient amount of iron can be administrated during preoperative. Currently, there is no evidence to elucidate whether short-term sufficient intravenous iron supplementation can reduce perioperative blood transfusion requirements among IDA patients. Thus, we hypothesized that short-term intravenous administration of sufficient iron isomaltose anhydride can reduce the need for perioperative allogeneic RBC transfusion without increasing the incidence of adverse reactions.

This prospective, randomized, controlled study aims to evaluate the impact of short-term (1 week) intravenous iron isomaltose anhydride in preoperative IDA patients receiving orthopedic surgery on postoperative allogeneic RBC transfusion rate and amount, hemoglobin level and iron storage, postoperative complications, average length/expense of hospital stay, etc., to determine the safety and efficacy of short-term sufficient intravenous iron therapy, and to develop a simple and effective preoperative iron supplementation program.

ELIGIBILITY:
Inclusion Criteria:

* Age > 14 years;
* Sign and date the "informed consent form"

Exclusion Criteria:

* Pregnant or lactation;
* Drug abuse, including but not limited to opioids, amphetamines, ice, ketamine, etc.;
* History of anaphylaxis to oral or intravenous iron;
* Nervous system diseases such as peripheral neuropathy, mental illness;
* Other conditions that the investigator deems are not suitable for the study, such as deafness, Parkinson's disease, communication disorders, etc.;
* Participated in other clinical trials during the first three months of the study.

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2024-07-05 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of allogeneic RBC transfusion | 30 days after randomization
  Number of patients who receive allogeneic RBC transfusion/total number of patients.

SECONDARY OUTCOMES:
Average number of units of RBC transfused in patients who receive allogeneic RBC transfusion | 30 days after randomization
  Total number of units of RBC transfused/number of patients who receive allogeneic RBC transfusion
Average number of units of RBC transfused in the entire study population | 30 days after randomization
  Total number of units of RBC transfused/total number of patients
Incidence of postoperative adverse events (AEs) | 30 days after randomization
  AEs are graded according to the severity:
  Grade 1 Recovery after temporary treatment, such as postoperative nausea and vomiting (PONV), urinary retention, anxiety, temporary insomnia, etc.
  Grade 2 Results in prolonged hospitalization, such as lung infections requiring antibiotic treatment, incision infections requiring debridement treatment, etc.; Grade 3 life-threatening, recovery after treatment during hospitalization, such as acute renal failure requiring renal replacement therapy, postoperative hemorrahge requiring surgical intervention, respiratory failure requiring mechanical ventilation, etc.; Grade 4 Injury last 30 days or more after surgery, a significant decrease in the quality of life, such as acute myocardial infarction, stroke, etc.; Grade 5 Death with 30 days after surgery
Hemoglobin (Hb) levels | 30 days after randomization
  Hemoglobin (Hb) levels at different time points;
Length of stay (LOS) | 30 days after randomization
  Length of stay (LOS), defined as number of days from admission to discharge
Postoperative hospital stay | 30 days after randomization
  Number of days from the day of surgery to discharge
Re-admission | 30 days after randomization
  Re-admission within 30 days after surgery
Cost of Hospitalization | 30 days after randomization
  Total cost of hospitalization from admission to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D., Principal Investigator — Department of Anesthesiology, West China Hospital, Sichuan University

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data could be accessed under request to Dr. Ren Liao by email: liaoren7733@163.com
Supporting Information: Study Protocol
Time Frame: From May 01,2023, for 10 years.
Access Criteria: Contact with Dr. Ren Liao by email: liaoren7733@163.com